CLINICAL TRIAL: NCT02056353
Title: LOGIC-Insulin Computerized Algorithm-guided Versus Nurse-directed Blood Glucose Control in Critically Ill Patients: the LOGIC-2 Multicentre Randomized Controlled Trial
Brief Title: Multicentre LOGIC-Insulin Algorithm-guided Versus Nurse-directed Blood Glucose Control During Critical Illness (LOGIC-2)
Acronym: LOGIC-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Principal Investigator, Greet Van den Berghe, Prof. Dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LOGIC-Insulin 2.1.1; ML9517 (Other: IRB-BE); S55613 (Other: University Hospitals Leuven); 80M0563 (Other: FAMHP); IWT-TBM 100793 (Other Grant/Funding Number: IWT-TBM)
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Critical Illness; Hyperglycemia; Hypoglycemia
Keywords: Software; Algorithm; Cardiac surgery
MeSH Terms: conditions — Critical Illness; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurse-directed (Active Comparator): Blood glucose control guided by paper protocol
  Interventions: Device: Paper protocol
- LOGIC-Insulin (Experimental): Blood glucose control guided by the LOGIC-Insulin algorithm
  Interventions: Device: LOGIC-Insulin algorithm

INTERVENTIONS:
Device: LOGIC-Insulin algorithm
  Arms: LOGIC-Insulin
Device: Paper protocol
  Arms: Nurse-directed

SUMMARY:
Most critically ill patients are confronted with hyperglycaemia, which is associated with an increased mortality and morbidity risk. Normalising these elevated blood glucose levels by intensive insulin therapy may improve patient outcome, but is associated with an increased risk of hypoglycaemia. The LOGIC-2 study hypothesises that the LOGIC-Insulin computerised software algorithm will allow better (less hyperglycaemia) and safer (less hypoglycaemia) blood glucose control in critically ill patients than nurse-directed blood glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU with an expected stay of at least 48 hours and already receiving or potentially needing insulin infusion for blood glucose control. These patients should already have or need an arterial and central venous line
* Patients should be 18 years or older

Exclusion Criteria:

* Not critically ill
* Age under 18 years
* Patients already enrolled in another intervention randomized controlled trial
* Patients expected to die within 12 hours (=moribund patients)
* No arterial line or central venous line needed
* Pregnancy or lactating
* Patients suffering from ketoacidotic or hyperosmolar coma on admission
* Patients who have been previously been included in the LOGIC-2 study
* Allergy to insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1550 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Glycemic Penalty Index (GPI) during the Intervention | up to 14 days post-randomization
  Adequacy of reaching and maintaining the target range for blood glucose during the intervention (Effectiveness of glycaemic control)

SECONDARY OUTCOMES:
Proportion of Patients With Severe Hypoglycaemia (<40 mg/dL) during the Intervention | up to 14 days post-randomization
  Proportion of patients to have had one or more episodes of severe hypoglycaemia (<40 mg/dL) during the intervention
Incidence of Severe Hypoglycemia (<40 mg/dL) during the Intervention | up to 14 days post-randomization
  Number of severe hypoglycaemic values as a fraction of all blood glucose measurements during the intervention
Blood Glucose Level Per Treatment Group during the Intervention | up to 14 days post-randomization
  Mean and median arterial blood glucose level
Hyperglycaemic index (HGI) | up to 14 days post-randomization
  Adequacy of reaching and maintaining the target range for blood glucose, as assessed by the Hyperglycaemic index (HGI)
Time in target range | up to 14 days post-randomization
Time to target range | up to 14 days post-randomization
Daily maximal blood glucose difference | up to 14 days post-randomization
  marker of blood glucose fluctuations
Incidence of mild hypoglycaemia (blood glucose level < 70 mg/dL or 3.9 mmol/L) during the Intervention | up to 14 days post-randomization
  Number of mild hypoglycaemic values as a fraction of all blood glucose measurements during the intervention
Proportion of Patients With Mild Hypoglycaemia (blood glucose level < 70 mg/dL or 3.9 mmol/L) during the Intervention | up to 14 days post-randomization
  Proportion of patients to have had one or more episodes of mild hypoglycaemia during the intervention
Interval between blood glucose measurements | up to 14 days post-randomization
  marker of workload
Protocol compliance in the intervention group | up to 14 days post-randomization
  the number and proportion of patients in which the LOGIC-Insulin was not followed for a time period of at least 8 hours, which is the duration of one nurse shift.
Overrules in the intervention group | up to 14 days post-randomization
  the number and proportions of recommendations by the software that were overruled by the bed-side nurses
  * Minor overrules: absolute insulin dose difference of >0.1 and < 1IU/h
  * Major overrules: absolute insulin dose difference of >= 1IU/h
  * Major overrules will also be qualitatively assessed
Incidence of new infections in the ICU | up to 90 days post-randomization
  The diagnosis of "new infection" will be based on the administration of antibiotics, beyond the prophylactic scope
Length of stay in the ICU | up to 90 days post-randomization
Length of stay in the hospital | up to 90 days post-randomization
Mortality in the ICU | up to 90 days post-randomization
Mortality in the hospital | up to 90 days post-randomization
Landmark 90-day mortality | up to 90 days post-randomization
All direct medical costs from a healthcare payer's perspective | up to 90 days post-randomization
Quality of Life | up to 90 days post-randomization
  EuroQol-5D

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Mesotten, MD, PhD, Study Director — KU Leuven; Greet Van den Berghe, MD, PhD, Principal Investigator — KU Leuven; Jasperina Dubois, MD, Principal Investigator — Jessa hospital, Hasselt; Marcus Schultz, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (4):
- Belgium (3):
  - Jessa Hospital, Hasselt
  - Dept Intensive Care Medicine, University Hospitals Leuven, Leuven
  - Medical Intensive Care, University Hospitals Leuven, Leuven
- Academic Medical Center (AMC), Amsterdam, Netherlands

REFERENCES:
- [Background] Van Herpe T, Mesotten D, Wouters PJ, Herbots J, Voets E, Buyens J, De Moor B, Van den Berghe G. LOGIC-insulin algorithm-guided versus nurse-directed blood glucose control during critical illness: the LOGIC-1 single-center, randomized, controlled clinical trial. Diabetes Care. 2013 Feb;36(2):188-94. doi: 10.2337/dc12-0584. Epub 2012 Sep 6. PMID 22961576
- [Background] Van Herpe T, De Brabanter J, Beullens M, De Moor B, Van den Berghe G. Glycemic penalty index for adequately assessing and comparing different blood glucose control algorithms. Crit Care. 2008;12(1):R24. doi: 10.1186/cc6800. Epub 2008 Feb 26. PMID 18302732
- [Background] Van den Berghe G, Schetz M, Vlasselaers D, Hermans G, Wilmer A, Bouillon R, Mesotten D. Clinical review: Intensive insulin therapy in critically ill patients: NICE-SUGAR or Leuven blood glucose target? J Clin Endocrinol Metab. 2009 Sep;94(9):3163-70. doi: 10.1210/jc.2009-0663. Epub 2009 Jun 16. PMID 19531590
- [Derived] Dubois J, Van Herpe T, van Hooijdonk RT, Wouters R, Coart D, Wouters P, Van Assche A, Veraghtert G, De Moor B, Wauters J, Wilmer A, Schultz MJ, Van den Berghe G, Mesotten D. Software-guided versus nurse-directed blood glucose control in critically ill patients: the LOGIC-2 multicenter randomized controlled clinical trial. Crit Care. 2017 Aug 14;21(1):212. doi: 10.1186/s13054-017-1799-6. PMID 28806982